CLINICAL TRIAL: NCT00044135
Title: A Phase II, Randomized, Partially-Blinded Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of 12 Weeks of Treatment with Clevudine (10 mg, 30 mg or 50 mg QD) in Patients Infected with Hepatitis B Virus.
Brief Title: A Safety Study to Evaluate 12 Weeks of Treatment with Clevudine in Patients Infected with Hepatitis B Virus.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Triangle Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-FMAU-102 B
Record Dates: First submitted 2002-08-20; First posted 2002-08-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-11

CONDITIONS: Hepatitis B
Keywords: clevudine; hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: clevudine (drug)

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of 12 weeks of treatment with clevudine, at one of three doses, in patients chronically infected with hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* HBV DNA positive with DNA levels at screening greater than or equal to 3,000,000 copies/mL.
* Documented to be HBsAg positive for > 6 months OR HBsAg positive and IgM anti-HBc negative and anti-HBs negative. Patients may be HBeAg positive, and anti-HBe negative OR HBeAg negative (pre-core mutant) and anti-HBe positive.
* HBeAg positive and anti-HBe negative OR HBeAg negative (pre-core mutant) and anti-HBe positive with positive HBsAg for the previous 6 months
* AST and ALT levels which are less than or equal to 10 times the upper limit of normal.
* Bilirubin levels less than or equal to 1.5 x ULN or bilirubin levels > 1.5 x ULN with diagnosis of Gilbert's disease and conjugated bilirubin within normal limits.

Exclusion Criteria:

* Currently receiving antiviral, immunomodulatory or corticosteroid therapy
* Previous treatment with lamivudine, lobucavir, adefovir, famciclovir, or any other investigational nucleoside for HBV infection
* Previous treatment with interferon must have ended at least 6 months prior to screening visit
* History of ascites, variceal hemorrhage or hepatic encephalopathy
* Co-infection with HCV or HIV
* Evidence of cirrhosis or hepatocellular carcinoma (alpha fetoprotein)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2002-08

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Thomas Jefferson University Hospital, Jefferson Medical College, Philadelphia, Pennsylvania
- Canada (2):
  - Viridae, Vancouver
  - University of British Columbia, Downtown Infectious Disease Clinic, Vancouver
- China (2):
  - Prince of Wales Hospital, Department of Medicine and Therapeutics, Hong Kong
  - The University of Hong Kong, Clinical Trials Centre, Faculty of Medicine, Queen Mary Hospital, Hong Kong
- France (4):
  - Hospital Beaujon, Service Hepatologie Centre Pierre Abrami, Clichy
  - Hospital Dieu, Service Hepatogastroenterologie-endoscopie, Lyon
  - Hospital St Louis, Service de Medecine Interne, Paris
  - Hospital de Brabois Chu de Nancy, Service d'Hepato-gastroenterologie, Vandœuvre-lès-Nancy
- National University Hospital, Division of Gastroenterology, Department of Medicine, Singapore, Singapore